CLINICAL TRIAL: NCT01177072
Title: Study of Effectiveness of Mental Health Interventions Among Torture Survivors in Southern Iraq
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Heartland Alliance (Other); Ministry of Health, Iraq (Network); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, William Weiss, Assistant Scientist, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JHSPH-3034
Record Dates: First submitted 2010-07-16; First posted 2010-08-06 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Depression; Anxiety; Post-Traumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Components-Based Interventions (CBI) (Experimental): 12 sessions of cognitive processing therapy. Sessions are expected to be approximately one week apart. Although each counseling session is designed to be carried out one week apart for a total of 12 weeks, there are many reasons why a session will be missed. Our estimation is that a single client will require 4-5 months to complete the therapy.
  Interventions: Other: Components-Based Intervention
- Cognitive Processing Therapy (Experimental): 12 sessions of cognitive processing therapy. Sessions are expected to be approximately one week apart. Although each counseling session is designed to be carried out one week apart for a total of 12 weeks, there are many reasons why a session will be missed. Our estimation is that a single client will require 4-5 months to complete the therapy.
  Interventions: Other: Cognitive Processing Therapy
- Wait List Control (No Intervention): Eligible clients will not be provided therapy at enrollment. After the study period has completed, control clients will be re-interviewed. Those that remain eligible due to symptom cutoff scores will be offered therapy. In the interim, controls will receive a phone call once a month; those with indications of possible harm to self or others will be referred to a psychiatrist.

INTERVENTIONS:
Other: Cognitive Processing Therapy — 12 sessions of cognitive processing therapy. Sessions are expected to be approximately one week apart. Although each counseling session is designed to be carried out one week apart for a total of 12 weeks, there are many reasons why a session will be missed. Our estimation is that a single client will require 4-5 months to complete the therapy.
  Arms: Cognitive Processing Therapy
Other: Components-Based Intervention — This is a 'components-based' intervention include psychoeducation, relaxation, life-enhancing skills (problems solving and safety planning), exposure, and cognitive processing of life problems and traumatic events. The duration of sessions are approximately one hour), the expected frequency of treatment is weekly, and recommended number of sessions are 12.
  Arms: Components-Based Interventions (CBI)

SUMMARY:
1. That the psychotherapeutic intervention - Components-Base Interventions (CBI) - is effective in reducing the severity of mental health symptoms experienced by torture survivors in Southern Iraq.
2. That the psychotherapeutic intervention - Cognitive Processing Therapy (CPT) - is effective in reducing the severity of mental health symptoms experienced by torture survivors in Southern Iraq.

DETAILED DESCRIPTION:
For each intervention, participants will undergo 12 sessions (CBI or CPT) that are standardized by training and manual for community mental health workers (CHMWs). CMHWs will be trained in only one intervention. Prior to the starting sessions, a baseline assessment of depression, anxiety and trauma symptoms and function will be carried out. A follow up assessment will be carried out after the 12 sessions have been completed. Expected time between sessions is one week. The total time per client is expected to last about 4-5 months to complete the 12 therapy sessions.

Participants will be randomized (within CMHW) to either immediate intervention or wait-list control. Participants that are wait-list control will be contacted monthly for assessment of condition. Any participant (intervention or control) with suicidal thoughts or distress that does not abate will be referred for psychiatric care.

ELIGIBILITY:
Inclusion Criteria:

* Exposure to Torture
* PTSD

Exclusion Criteria:

* Children
* Mentally incompetent to understand therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Severity of Trauma. This will be the difference in group mean score of severity of depression based on a sum of ratings of various standard depression symptoms from the Hopkins Symptom Checklist and locally defined symptoms. | After 12 counseling , 4-5 months
  Although each counseling session is designed to be carried out one week apart for a total of 12 weeks, there are many reasons why a session will be missed. Our estimation is that a single client will require 4-5 months to complete the therapy.

SECONDARY OUTCOMES:
Ability to Function. This is the difference in group mean of ability to function based on the sum of ratings of functional ability among various tasks identified by the local population as important functions (men and women have separate tasks). | After 12 counseling session, estimated 4-5 months.
  Although each counseling session is designed to be carried out one week apart for a total of 12 weeks, there are many reasons why a session will be missed. Our estimation is that a single client will require 4-5 months to complete the therapy.

CONTACTS AND LOCATIONS:
Overall Officials: William M Weiss, DrPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Ministry of Health Iraq, Several Cities in Iraq (Karbala, Basra, Najaf, Etc.), Iraq

REFERENCES:
- [Derived] Weiss WM, Murray LK, Zangana GA, Mahmooth Z, Kaysen D, Dorsey S, Lindgren K, Gross A, Murray SM, Bass JK, Bolton P. Community-based mental health treatments for survivors of torture and militant attacks in Southern Iraq: a randomized control trial. BMC Psychiatry. 2015 Oct 14;15:249. doi: 10.1186/s12888-015-0622-7. PMID 26467303